CLINICAL TRIAL: NCT03700099
Title: Prospective Biomarker Analysis of Patients With Metastatic Castration-resistant Prostate Cancer (mCRPC) Undergoing Sequential Treatment With Docetaxel and Enzalutamide
Brief Title: Biomarker Analysis of Castration-resistant Prostate Cancer Undergoing Treatment With Docetaxel Followed by Enzalutamide
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 1082/17
Record Dates: First submitted 2018-09-14; First posted 2018-10-09 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer; Castration-resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Drug Therapy; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study cohort (Other): Docetaxel 75 mg/m2 i.v. every 3 weeks for 6-10 cycles. Upon disease progression after docetaxel, participants will receive enzalutamide 160 mg p.o. daily until limiting toxicity or disease progression.
  Interventions: Drug: Docetaxel; Drug: Enzalutamide

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/m2 IV every 3 weeks, for 6-10 cycles.
  Other Names: Chemotherapy
Drug: Enzalutamide — Upon disease progression after treatment with docetaxel, patients will receive Enzalutamide 160 mg P.O. daily until disease progression or limiting toxicity.
  Other Names: Xtandi

SUMMARY:
This is a prospective biomarker study of patients with metastatic castration-resistant prostate cancer (mCRPC) undergoing sequential treatment with docetaxel and enzalutamide. The participants will undergo serial pre- and post-therapy blood collection for biomarker analysis as part of the primary objective of the study. The primary goal of this study is to evaluate the association of the AR-V7 status and androgen receptor (AR) gene alterations with PSA response to docetaxel and enzalutamide.

DETAILED DESCRIPTION:
This study is a prospective biomarker study of patients with metastatic castration-resistant prostate cancer (mCRPC) undergoing sequential treatment with docetaxel followed by enzalutamide. In this study, all participants will receive standard of care treatment with docetaxel 75 mg/m2 every 3 weeks up to 10 cycles and after progression, patients will receive enzalutamide 160 mg daily until limiting toxicity or disease progression. The participants will undergo serial pre- and post-therapy blood collection for biomarker analysis as part of the primary objective of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Men diagnosed with metastatic prostate cancer, with at least one metastatic lesion on CT or bone scan.
* Documentation of castrate levels of testosterone (< 50 ng per deciliter), and continued androgen deprivation therapy or surgical castration.
* Progressive disease at study entry defined as one or more of the following three criteria that occurred while the patient was on androgen deprivation therapy:

  * PSA progression defined by a minimum of two rising PSA levels with an interval of ≥

    1 week between each determination. Patients who received an anti-androgen must have progression after withdrawal (≥ 4 weeks since last flutamide, bicalutamide or nilutamide). The PSA value at the Screening visit should be ≥ 2 μg/L (2 ng/mL);
  * Soft tissue disease progression defined by RECIST 1.1;
  * Bone disease progression defined by PCWG2 with two or more new lesions on bone scan.
* No prior chemotherapy for mCRPC.
* Patients previously treated with bicalutamide, ketoconazole, or estrogens will be eligible. These patients must have discontinued therapy ≥ 4 weeks prior to enrollment.
* Patients previously treated with steroids or receiving prednisone or dexamethasone will be eligible. In this case, continuing therapy will be at the discretion of the attending physician.
* Patients who are candidates for therapy with docetaxel and enzalutamide.
* Patients must agree to undergo pre- and post-therapy blood collection.
* Patients must understand and be willing to sign the written informed consent form of this study.

Exclusion Criteria:

* Patients with CRPC previously treated with chemotherapy.
* Non-castrate levels of testosterone (> 50 ng per deciliter) or inability to continue androgen deprivation therapy during the study period.
* Absence of detectable metastasis on imaging studies.
* Prior therapy with abiraterone, enzalutamide or any investigational AR-directed agent.
* Contra-indication for therapy with docetaxel or enzalutamide.
* History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke or significant brain trauma). History of loss of consciousness or transient ischemic attack within 12 months of enrollment.
* Known or suspected brain metastasis or active leptomeningeal disease.
* Severe concurrent disease, infection, or co-morbidity that, in the judgment of the Investigator, would make the patient inappropriate for enrollment;
* History of another malignancy within the previous 5 years other than curatively treated non-melanomatous skin cancer;
* Absolute neutrophil count < 1,500/μL, or platelet count < 100,000/μL, or hemoglobin < 9 g/dL at the Screening visit;
* Total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal at the screening visit (for Docetaxel phase only);
* Creatinine > 2 mg/dL at the Screening visit (for Docetaxel phase only);
* Albumin < 3.0 g/dL at the Screening visit (for Docetaxel phase only);
* Clinically significant cardiovascular disease including:

  * Myocardial infarction within 6 months;
  * Uncontrolled angina within 3 months;
  * Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or patients with history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multi-gated acquisition scan performed within three months results in a left ventricular ejection fraction that is ≥ 45%;
* History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes);
* History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place;
* Hypotension as indicated by systolic blood pressure < 86 millimeters of mercury (mmHg) at the screening visit;
* Bradycardia as indicated by a heart rate of < 50 beats per minute on the Screening ECG;
* Uncontrolled hypertension as indicated by systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg at the Screening visit;
* Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease within last 3 months);
* Major surgery within 4 weeks of enrollment (Day 1 Visit);
* Radiation therapy for treatment of the primary tumor within 3 weeks of enrollment (Day 1 visit);
* Treatment with flutamide, bicalutamide or nilutamide within 4 weeks of enrollment (Day 1 visit);
* Treatment with 5-α reductase inhibitors (finasteride, dutasteride), estrogens, cytproterone within 4 weeks of enrollment (Day 1 visit)
* Treatment with systemic biologic therapy for prostate cancer (other than approved bone targeted agents and GnRH analogue therapy) or other agents with anti-tumor activity within 4 weeks of enrollment (Day 1 visit);
* Prior use, or participation in a clinical trial, of an investigational agent that blocks androgen synthesis (e.g., abiraterone acetate, TAK-700) or targets the androgen receptor, including enzalutamide.
* Use of an investigational agent within 4 weeks of enrollment (Day 1 visit);
* Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of 10 mg of prednisone per day within four weeks of enrollment (Day 1 visit);
* Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of safety data;
* Participation in a previous clinical trial of enzalutamide or an investigational agent that inhibits the androgen receptor or androgen synthesis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Correlate AR-V7 status in circulating tumor cells (positive versus negative) and PSA response decline > 50% after therapy with docetaxel | 6 months
Correlate AR-V7 status in circulating tumor cells (positive versus negative) and PSA decline > 50% after therapy with enzalutamide | 12 months
Correlate AR mutations (present versus absent) and PSA response decline > 50% after therapy with docetaxel. | 6 months
Correlate AR mutations (present versus absent) and PSA response decline > 50% after therapy with enzalutamide. | 12 months

SECONDARY OUTCOMES:
Correlate AR-V7 status in circulating tumor cells (positive versus negative) and time to PSA progression after docetaxel. | 12 months
Correlate AR-V7 status in circulating tumor cells (positive versus negative) and time to PSA progression after enzalutamide. | 12 months
Correlate AR mutations (present versus absent) and time to PSA progression after docetaxel. | 12 months
Correlate AR mutations (present versus absent) and time to PSA progression after enzalutamide. | 12 months
Correlate AR-V7 status in circulating tumor cells (positive versus negative) and overall survival. | 24 months
Correlate AR mutations (present versus absent) and median overall survival. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Diogo Bastos, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No